CLINICAL TRIAL: NCT07000890
Title: Rheumatoid Arthritis Synovial Tissue Biopsy Study
Acronym: RAST-BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/28AVR/252
Record Dates: First submitted 2022-06-20; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Synovial biopsy (Experimental): Assessment of the effects of TNF blockade on cells isolated from RA synovial tissue prior to and 12 weeks after initiation of therapy.
  Interventions: Diagnostic Test: Synovial Biopsy

INTERVENTIONS:
Diagnostic Test: Synovial Biopsy — Synovial tissue and blood samples will be collected and processed for bulk and scRNAseq; serum, plasma, DNA, RNA and PBMCs as per below flow chart. Biomarker exploratory analysis will be performed.

SUMMARY:
In this proof-of-concept study, the investigators intend to collect synovial biopsies from MTX-resistant RA patients prior to and 12 weeks after initiation of TNF-blocking therapy (period 1). In addition to conventional histological and immunohistochemistry characterization of the samples, single cell RNASeq studies will be performed, with a particular focus on synovial T cells and fibroblasts. Clinical response to TNF blocking therapies will be assessed using validated measurements, which will result in the identification of novel mechanisms and markers of resistance to TNF inhibition in MTX-resistant RA patients.

DETAILED DESCRIPTION:
All patients (n=50) included in this trial will be diagnosed with RA according to the ACR/EULAR 2010 classification criteria. They will be eligible for standard-of-care therapy using TNF blockers, because they have active disease despite previous administration of two conventional DMARDs (including methotrexate) for a period of at least 3 months each. Disease activity at study entry (before initiation of TNF blockade) and at 12 weeks will be assessed using DAS28-CRP (composite score that integrates numbers of tender and swollen joints, serum CRP concentrations, and patient's evaluation of disease activity on a visual analogic scale) and EULAR response criteria. All treatments other than TNF blockade will be stable for at least 4 weeks before study entry, and for the whole duration of the study (4 months after initiation of TNF blockade). All clinical assessments will be performed by the investigators.

Efficacy will be assessed according to the ACR/EULAR core set of response (DAS28-CRP, CDAI, SDAI, HAQ) of TNFi and JAKi in period 2 for non-responders to TNFi.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females (not nursing and not pregnant) at least 18 years of age. Women of child-bearing potential are eligible if they are practicing effective contraceptive measures.
2. Subjects must meet the criteria of the 2010 EULAR/ACR criteria for the diagnosis of rheumatoid arthritis
3. Subjects must have a disease activity as defined by a tender joint count > 4, swollen joint count > 4 from 68 joints and a DAS28-CRP >3.7. (This value is the cut off level to obtain a reimbursement for bDMARDs in Belgium).
4. Subjects were treated with MTX 15 mg a week (or 7.5 mg in case of poor tolerance) for at least 3 months.
5. Subjects must be naive to TNF inhibitors (Adalimumab, Etanercept, Infliximab, Certolizumab, Golimumab) and other b- or tsDMARDs (Abatacept, Tocilizumab, Rituximab and JAK inhibitors)

Exclusion Criteria:

1. Women of child-bearing age who are unwilling or unable to use an acceptable method to avoid pregnancy
2. Women who are pregnant or breastfeeding
3. Subjects with a history of cancer within the last five years (other than nonmelanoma skin cell cancers cured by local resection). Existing non-melanoma skin cell cancers must be removed prior to dosing.
4. Subjects with any serious bacterial infection and at risk for tuberculosis (TB).
5. Subjects who are unable to accept and perform the synovial biopsy procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Primary resistance to TNF blockade in synovium | 6 months
  Identification of novel mechanisms associated with primary resistance to TNF blockade in synovial biopsies using single cell RNASeq analyses

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, Principal Investigator — UCLouvain - IREC
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No